CLINICAL TRIAL: NCT04202172
Title: Six-month Endothelial and Microcirculatory Function of the Bioactive Sirolimus-eluting Combo Stent Versus the Polymer-free Biolimus-eluting Biofreedom Stent in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Functional Assessment of the Infart-related Artery With Bioactive and Polymer-free Coronary Stents (The FUNCOMBO Trial)
Acronym: FUNCOMBO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Josep Gomez Lara, Principal Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC009/18
Record Dates: First submitted 2018-10-28; First posted 2019-12-17 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Endothelial Dysfunction; Coronary Microvascular Disease; Myocardial Infarction
Keywords: endothelial function
MeSH Terms: conditions — Microvascular Angina; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BIOFREEDOM (Active Comparator): Implantation of Drug-eluting coronary stent without polymer in patients with myocardial infarction.
  Interventions: Procedure: Stent implantation in the infart-related artery in patients with ST elevation myocardial infarction
- COMBO (Experimental): Implantation of Bioactive coronary stent in patients with myocardial infarction.
  Interventions: Procedure: Stent implantation in the infart-related artery in patients with ST elevation myocardial infarction

INTERVENTIONS:
Procedure: Stent implantation in the infart-related artery in patients with ST elevation myocardial infarction — The 6-month scheduled coronary angiography will perform 3 interventions:
  1. Endothelial function assessment with intracoronary acetyl-choline infusion.
  2. Microcirculatory function assessment with a pressure wire during endovenous adenosine infusion.
  3. Stent healing assessment using optical coherence tomography
  Other Names: All patients will undergo to 6-month coronary angiography after stent implantation in order to assess the endothelial and microvascular function of the infarct related artery

SUMMARY:
A total of 50 patients with ST-elevation myocardial infarction (STEMI) undergoing primary-percutaneous coronary intervention (PPCI) will be randomized to two different coronary stents: BIOFREEDOM vs. COMBO stent.

All patients will undergo to 6-month scheduled coronary angiography to evaluate the endothelial function response of the distal coronary segment and other functional parameters.

DETAILED DESCRIPTION:
The bioengineered COMBO stent (Orbus Neich, Fort Lauderdale, Florida, United States) has a dual-therapy strategy, which combines a sirolimus-eluting coating with an anti-CD34 antibody layer to promote vessel healing. Sirolimus release (5 μg/mm) is completed in 30 days, and the biodegradable polymer disappears within 90 days.

CD34 antibodies are immobilized on the surface of the stent and capture circulating endothelial progenitor cells (EPCs). The captured EPCs are triggered by sheer stress from the circulating blood and other cell signals to differentiate and mature into endothelial cells. COMBO Plus is the only stent with a biological coating that actively repairs the vessel morphology. However, little is known regarding the endothelial function after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* STEMI < 12 hours undergoing primary PCI.
* ST-segment elevation of > 1mm in > 2 contiguous leads, or (presumably new) left bundle branch block, or true posterior MI with ST depression of >1mm in >2 contiguous anterior leads.
* Presence of at least one acute infarct artery target vessel with one or more de-novo coronary artery stenosis in a native coronary artery within 2.75 - 3.75 mm reference vessel diameter and < 24 mm length (visually estimated).

Exclusion Criteria:

* Inability to provide informed consent
* Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy
* Known intolerance to aspirin, heparin, PLLA, everolimus, contrast material
* Cardiogenic Shock
* Unprotected left main coronary artery stenosis
* Distal occlusion of target vessel
* Acute myocardial infarction secondary to stent thrombosis
* Mechanical complications of acute myocardial infarction
* Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in sub-optimal imaging or excessive risk of complication in the follow-up procedure
* Active bleeding or coagulopathy or patients at chronic anticoagulation therapy
* Chronic renal dysfunction with creatinine clearance < 45 ml/minm2
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function of the distal coronary segment of patients with myocardial infarction treated with two types of drug-eluting stents | At 6 months of the stent implantation
  To compare the mean lumen diameter changes to intracoronary acetyl-choline infusion of the distal coronary segment by quantitative coronary angiography between the COMBO stent vs. the BIOFREEDOM stent in STEMI patients. Endothelial dysfunction is defined as >4% vasoconstriction to intracoronary acetylcholine compared to the 6-month baseline mean lumen diameter of the matched segment.

SECONDARY OUTCOMES:
Index of microcirculatory resistance | At 6 months of the stent implantation
  To compare the index of microcirculatory resistance (IMR) between the culprit arteries treated with COMBO vs. BIOFREEDOM in STEMI patients.
Coronary flow reserve | At 6 months of the stent implantation
  To compare the coronary flow reserve (CFR) between the culprit arteries treated with COMBO vs. BIOFREEDOM in STEMI patients

OTHER OUTCOMES:
Fractional flow reserve | At 6 months of the stent implantation
  To compare the fractional flow reserve (FFR) between the culprit arteries treated with COMBO vs. BIOFREEDOM in STEMI patients

CONTACTS AND LOCATIONS:
Overall Officials: Josep Gomez Lara, MD PhD, Principal Investigator — Hospital Universitari de Bellvitge, L´Hospitalet de Llobregat, Spain; Neus Salvatella, MD, Principal Investigator — Hospital del Mar, Barcelona, Spain; Salvatore Brugaletta, MD PhD, Principal Investigator — Hospital Clinic, Barcelona, Spain
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez-Lara J, Oyarzabal L, Brugaletta S, Salvatella N, Romaguera R, Roura G, Fuentes L, Perez Fuentes P, Ortega-Paz L, Ferreiro JL, Teruel L, Gracida M, Vaquerizo B, Sabate M, Comin-Colet J, Gomez-Hospital JA. Coronary endothelial and microvascular function distal to polymer-free and endothelial cell-capturing drug-eluting stents. The randomized FUNCOMBO trial. Rev Esp Cardiol (Engl Ed). 2021 Dec;74(12):1013-1022. doi: 10.1016/j.rec.2021.01.007. Epub 2021 Feb 24. English, Spanish. PMID 33640311